CLINICAL TRIAL: NCT02530021
Title: Sixty Minutes Heart Rate Variability Testing Compared With Non-invasive Exercise Stress Test in Hospitalized Patients With Suspected Angina Pectoris
Brief Title: Heart Rate Variability (HRV) Testing Compared With Exercise Stress Test in Hospitalized Patients With Chest Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Arnson Yoav, Dr., Meir Medical Center
Other Study IDs: 0036-15
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Angina Pectoris; Ischemic Heart Disease
Keywords: Ischemic heart disease; Heart rate variability; Exercise Strss Test
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart rate monitor: Hospitalized patients with chest pain and suspected ischemic heart disease who are candidates for non invasive exercise stress test by their treating physician.
  The patients will perform a one hour heart rate variability monitoring prior to the stress test.
  Interventions: Other: Heart rate monitor

INTERVENTIONS:
Other: Heart rate monitor — One hour non-invasive ECG heart rate variability monitoring. The results will be blinded and interpreted independantly. Study results will not effect patient management.

SUMMARY:
There are many patients hospitalized for chest pain, which don't have high risk features that require invasive coronary angiography, but are considered intermediate risk and for which ischemic heart disease can not be excluded.

The current management for these patients is to perform a non invasive test in order to classify their risk.

Exercise ergometry is a commonly used non invasive test to detect ischemia. that test is non-invasive, and does not involve radiation or intra-venous contrast. The test is limited for many patients, because of un-ability to exercise, or because of non-interpetable Electro Cardio-Graphy (ECG).

Heart rate variability is well known to be a marker of ischemic heart disease. Heart rate variability testing is a non-invasive ECG monitoring technique.

The study design is to identify hospitalized patients who are candidates for non-invasive stress testing, and to monitor their heart rate variability for one hour prior to the stress test.

DETAILED DESCRIPTION:
Ischemic heart disease is among the leading causes of death and disability in the modern world. Effective treatment for cardiac ischemia is based on identification of the proper patients and assigning prompt treatment to those patients.

It is not simple identifying the proper patients. There are many patients complaining of typical anginal chest pain without coronary heart disease, and there are many patients with active angina who complain of non-typical symptoms or who don't feel any symptoms.

Management of hospitalized patients with suspected angina pectoris is based on their complaints, their risk factors and laboratory results (ECG, troponin). They are classified into low-risk, high risk and intermediate.

Intermediate risk patients usually require additional testing in the hospital in order to re-classify them into high or low risk.

Heart rate variability is a well-known marker of active cardiac ischemia. The investigators plan to perform a 60 minute heart rate variability monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Hospitalized for Chest pain
* Intermediate probability for ischemic heart disease
* Selected management strategy is non invasive cardiac stress testing

Exclusion Criteria:

* Active Ischemic symptoms
* ECG changes suggestive of myocardial ischemia
* Troponin elevation on blood tests
* Atrial flutter
* Multiple APB's or VPB's on resting ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with suspected ischemic heart disease requiring further evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Correlation betwen Heart rate variability test and non-onvasive testing | The time from non-invasive testing to hospital discharg. Estimated up to 5 Days
  Heart rate variability results will be compared to non-invasive test results ordered as routine care by treating physician.

SECONDARY OUTCOMES:
Correlation between Heart rate variability and invasive angiography | Time from non-invasive testing to coronary angiography. Estimated up to 5 days
  Patients which will undergo invasive angiography as part of selected management strategy will be compared with Heart rate variability test results.

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Arnson, MD, Principal Investigator — Mei Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Harris PR, Stein PK, Fung GL, Drew BJ. Heart rate variability measured early in patients with evolving acute coronary syndrome and 1-year outcomes of rehospitalization and mortality. Vasc Health Risk Manag. 2014 Aug 5;10:451-64. doi: 10.2147/VHRM.S57524. eCollection 2014. PMID 25143740